CLINICAL TRIAL: NCT02601703
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multiple-Site Study to Evaluate the Therapeutic Equivalence of a Generic Tacrolimus Ointment, 0.1% (Glenmark Pharmaceuticals, Ltd) to the Marketed Product Protopic® (Tacrolimus) Ointment, 0.1% (Astellas Pharma US, Inc.) in the Treatment of Moderate to Severe Atopic Dermatitis (AD)
Brief Title: To Study Generic Tacrolimus Ointment, 0.1% in the Treatment of Moderate to Severe Atopic Dermatitis (Inflammation of Skin: Itchy, Red, Swollen, and Cracked Skin)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GLK-1501
Record Dates: First submitted 2015-11-09; First posted 2015-11-10 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tacrolimus Ointment 0.1% (Experimental)
  Interventions: Drug: Tacrolimus Ointment 0.1%
- Protopic® ointment, 0.1% (Active Comparator)
  Interventions: Drug: Protopic® ointment, 0.1%
- Placebo of Tacrolimus Ointment (Placebo Comparator)
  Interventions: Drug: Placebo of Tacrolimus Ointment

INTERVENTIONS:
Drug: Tacrolimus Ointment 0.1% — apply thin layer of ointment to affected area
  Arms: Tacrolimus Ointment 0.1%
Drug: Protopic® ointment, 0.1% — apply thin layer of ointment to affected area
  Arms: Protopic® ointment, 0.1%
Drug: Placebo of Tacrolimus Ointment — apply thin layer of ointment to affected area
  Arms: Placebo of Tacrolimus Ointment

SUMMARY:
This is a Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multiple-Site Study to Evaluate the Therapeutic Equivalence of a Generic Tacrolimus Ointment, 0.1% (Glenmark Pharmaceuticals, Ltd) to the Marketed Product Protopic® (tacrolimus) ointment, 0.1% (Astellas Pharma US, Inc.) in the Treatment of Moderate to Severe Atopic Dermatitis (AD).

ELIGIBILITY:
Key Inclusion Criteria:

1. Non-immunocompromised male or non-pregnant, non-lactating female, 18 years of age or older with a clinical diagnosis of moderate to severe AD.
2. Have confirmed diagnosis of atopic dermatitis for at least 3 months using the diagnostic features as described by Hanifin and Rajka
3. Have an IGA score of 3 (moderate) or 4 (severe).
4. Have an affected Body Surface Area (BSA) of at least 20% at baseline.
5. Treated with a bland emollient for at least 7 days.

Key Exclusion Criteria:

1. Active cutaneous bacterial or viral infection in any treatment area at baseline.
2. Sunburn, extensive scarring, or pigmented lesion(s) in any treatment area at baseline.
3. History of confounding skin conditions, e.g., psoriasis, rosacea, erythroderma, or ichthyosis.
4. History or presence of Netherton's Syndrome, immunological deficiencies or diseases, HIV, diabetes, malignancy, serious active or recurrent infection, clinically significant severe renal insufficiency or severe hepatic disorders.
5. Known allergy or hypersensitivity to tacrolimus or any other component of the Study products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1110 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment (IGA) score of 0 or 1 within all treatment areas at the end of treatment | Day 15

SECONDARY OUTCOMES:
The change in severity score from baseline to study Day 15 of the four individual signs and symptoms of AD (i.e., erythema, induration/papulation, lichenification and pruritus). | Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nikhil Sawant, Study Director — Glenmark Pharmaceuticals Ltd
Locations (60):
- United States (60):
  - Glenmark Investigational Site 49, Tempe, Arizona
  - Glenmark Investigational Site 31, Anaheim, California
  - Glenmark Investigational Site 23, Bell Gardens, California
  - Glenmark Investigational Site 30, Cerritos, California
  - Glenmark Investigational Site 15, Chula Vista, California
  - Glenmark Investigational Site 14, La Mesa, California
  - Glenmark Investigational Site 1, Long Beach, California
  - Glenmark Investigational Site 17, Oceanside, California
  - Glenmark Investigational Site 25, Pasadena, California
  - Glenmark Investigational Site 20, San Ramon, California
  - Glenmark Investigational Site 44, Santa Ana, California
  - Glenmark Investigational Site 45, Brooksville, Florida
  - Glenmark Investigational Site 43, Coral Gables, Florida
  - Glenmark Investigational Site 34, Doral, Florida
  - Glenmark Investigational Site 22, Fort Lauderdale, Florida
  - Glenmark Investigational Site 35, Hialeah, Florida
  - Glenmark Investigational Site 59, Hialeah Gardens, Florida
  - Glenmark Investigational Site 11, Miami, Florida
  - Glenmark Investigational Site 19, Miami, Florida
  - Glenmark Investigational Site 33, Miami, Florida
  - Glenmark Investigational Site 40, Miami, Florida
  - Glenmark Investigational Site 42, Miami, Florida
  - Glenmark Investigational Site 50, Miami, Florida
  - Glenmark Investigational Site 51, Miami, Florida
  - Glenmark Investigational Site 54, Miami, Florida
  - Glenmark Investigational Site 56, Miami, Florida
  - Glenmark Investigational Site 58, Miami, Florida
  - Glenmark Investigational Site7, Miami, Florida
  - Glenmark Investigational Site 28, Miami Gardens, Florida
  - Glenmark Investigational Site 29, Miami Lakes, Florida
  - Glenmark Investigational Site 18, Miramar, Florida
  - Glenmark Investigational Site 32, North Miami Beach, Florida
  - Glenmark Investigational Site 48, Orlando, Florida
  - Glenmark Investigational Site 4, Ormond Beach, Florida
  - Glenmark Investigational Site 47, Pembroke Pines, Florida
  - Glenmark Investigational Site 5, Winter Park, Florida
  - Glenmark Investigational Site 52, Macon, Georgia
  - Glenmark Investigational Site12, Madisonville, Kentucky
  - Glenmark Investigational Site 2, Saint Joseph, Missouri
  - Glenmark Investigational Site 41, Henderson, Nevada
  - Glenmark Investigational Site 16, Las Vegas, Nevada
  - Glenmark Investigational Site 9, High Point, North Carolina
  - Glenmark Investigational Site 46, Wilmington, North Carolina
  - Glenmark Investigational Site 53, Cincinnati, Ohio
  - Glenmark Investigational Site 21, Cleveland, Ohio
  - Glenmark Investigational Site 36, Toledo, Ohio
  - Glenmark Investigational Site 3, Hazleton, Pennsylvania
  - Glenmark Investigational Site 57, West Columbia, South Carolina
  - Glenmark Investigational Site 6, Nashville, Tennessee
  - Glenmark Investigational Site 60, Baytown, Texas
  - Glenmark Investigational Site 27, Houston, Texas
  - Glenmark Investigational Site 39, Houston, Texas
  - Glenmark Investigational Site 8, Houston, Texas
  - Glenmark Investigational Site 24, Lampasas, Texas
  - Glenmark Investigational Site 37, Missouri City, Texas
  - Glenmark Investigational Site 10, Pflugerville, Texas
  - Glenmark Investigational Site 13, San Antonio, Texas
  - Glenmark Investigational Site 26, San Antonio, Texas
  - Glenmark Investigational Site 55, San Antonio, Texas
  - Glenmark Investigational Site 38, Sugar Land, Texas